CLINICAL TRIAL: NCT04655599
Title: Effect of Olorinab on Gastrointestinal Transit in Patients With Irritable Bowel Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: APD371-106
Record Dates: First submitted 2020-11-19; First posted 2020-12-07 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Olorinab; APD371; Irritable bowel syndrome; IBS; IBS with predominant constipation; IBS-C; IBS with predominant diarrhea; IBS-D
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — olorinab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olorinab, Then Placebo (Experimental): Participants will first receive olorinab, followed by a washout period, and they then will receive placebo.
  Interventions: Drug: Olorinab; Drug: Placebo
- Placebo, Then Olorinab (Placebo Comparator): Participants will first receive placebo, followed by a washout period, and they then will receive olorinab.
  Interventions: Drug: Olorinab; Drug: Placebo

INTERVENTIONS:
Drug: Olorinab — Olorinab tablet by mouth, 3 times a day for 4 days with a final dose on Day 5.
Drug: Placebo — Olorinab matching placebo tablet by mouth, 3 times a day for 4 days with a final dose on Day 5.

SUMMARY:
A Phase 1b study to determine the effect of oral olorinab on gastrointestinal transit in adult participants with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
This is a single-center, randomized, crossover, double-blind, placebo-controlled study designed to evaluate the effects of olorinab on gastric, small-bowel, and colonic transit in IBS participants with predominant constipation (IBS-C) or with predominant diarrhea (IBS-D).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of irritable bowel syndrome (IBS) with predominant constipation (IBS-C) or IBS with predominant diarrhea (IBS-D) according to Rome IV criteria at Screening
* Body mass index (BMI) 18.0 to 40.0 kilograms per square meter (kg/m^2), inclusive at Screening
* Negative test results for alcohol and selected drugs at Screening and Day 1
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative for human immunodeficiency virus (HIV) antibody screens at Screening
* Participants with recent (within 6 months of Screening) or ongoing alarm features (unexplained weight loss, nocturnal symptoms, blood mixed with stool) are to have had a diagnostic colonoscopy prior to Screening and after the onset of alarm features (for participants with alarm features) to exclude non-IBS conditions per the Rome IV diagnostic algorithm for IBS

Exclusion Criteria:

* Pregnant or lactating
* Structural or metabolic diseases/conditions that affect the gastrointestinal system
* Diagnosis of IBS with mixed bowel habits (IBS-M) or unsubtyped IBS (IBS-U)
* Unable to withdraw medications that alter gastrointestinal (GI) transit for 72 hours prior to baseline colonic transit assay through the duration of treatment period, with the exception of rescue medicine usage (bisacodyl and loperamide)
* Clinically relevant changes in dietary, lifestyle, or exercise regimen within 30 days prior to Screening and for the duration of the study that may confound efficacy assessments in the clinical judgment of the Investigator (or designee)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Colonic transit geometric center after consumption of radiolabeled meal, based on the delivery of activated charcoal in a methacrylate-coated capsule | up to 24 hours 30 minutes after consumption of radiolabeled meal
Gastric emptying half-life (t½) as determined by scintigraphic imaging of radiolabeled meal | up to 4 hours 10 minutes after consumption of radiolabeled meal

SECONDARY OUTCOMES:
Colonic transit geometric center after consumption of radiolabeled meal, based on the delivery of activated charcoal in a methacrylate-coated capsule | up to 48 hours 30 minutes after consumption of radiolabeled meal
Ascending colon emptying t½ of radiolabeled activated charcoal particles delivered in a methacrylate-coated capsule | up to 24 hours 30 minutes after consumption of radiolabeled meal
Gastric emptying after radiolabeled meal | at 2 hours ± 10 minutes and 4 hours ± 10 minutes after consumption of radiolabeled meal
Number and severity of adverse events | Up to approximately 6 weeks
  Safety will be assessed by monitoring adverse events and clinically relevant changes in vital signs and clinical laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No